CLINICAL TRIAL: NCT05210257
Title: Pain Education Added to Conventional Physiotherapy Program for Patients With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Özden YAŞARER, Principal investigator, Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ozdenyasarer neck pain
Record Dates: First submitted 2021-12-07; First posted 2022-01-27 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Neck Pain; Pain
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physiotherapy (Other): Conventional physiotherapy program consists of neck isometric exercises, neck isotonic exercises, stabilization exercises, stretching exercises and posture exercises and physiotherapy agents.
  Interventions: Other: Conventional physiotherapy
- Neuroscience education (Active Comparator): Conventional physiotherapy program and The neuroscience education trainings will be conducted in the form of face-to-face interviews and 45-50 minute one-to-one sessions.
  Interventions: Other: Neuroscience education

INTERVENTIONS:
Other: Conventional physiotherapy — Group 1 was given conventinal physiotherapy Physiotherapy agents; 5 min ultrasound 1.5 watts/cm2 20 min conventional TENS 20 min heat agent application (hot pack) Exercise program; Stretching and relaxation exercises, Neck strengthening exercises that include concentric and isometric contractions Posture exercises 3 sets per day, 1 in the hospital with 10 repetitions
  Arms: Conventional physiotherapy
Other: Neuroscience education — Conventional physiotherapy program and The neuroscience education trainings will be conducted in the form of face-to-face interviews and 45-50 minute one-to-one sessions.
  In sessions ; neurons and nerve conduction in the session, the formation process of pain, peripheral neuropathic pain, pain spread during the session, neuroplasticity, peripheral and central sensitization, hyperalgesia and allodynia, acute-chronic pain, The effects of stress, fear, anxiety, false thoughts and beliefs about pain and other psychosocial factors on the pain process and determining possible psychosocial factors in the patient during the session, Strategies for controlling the pain process and coping with psychosocial factors in the session will be completed by explaining the effect mechanisms of exercise on pain.
  Arms: Neuroscience education

SUMMARY:
Purpose: The aim of this study is to examine the effects of pain training applied with conventional physiotherapy on pain, range of motion, disability, kinesiophobia and quality of life in patients with neck pain.

Methods: The research is planned to be completed within 18 months at Istanbul Hospital.

It is planned to include 40 individualsbetween the ages of 18-65 with neck pain persisting for 3 months or more.Individuals will be randomly divided into 2 groups.

Conventional physiotherapy program will be applied to the first group. Conventional physiotherapy will be applied to the second group and neuroscience education will be given.Pain intensity will evaluate before and after exercise with 'Visual Analog Scale' (VAS), and algometer,range of motion will evaluate with C-ROM, kinesiofobia will questioned with Tampa Kinesiofobia Score, Quality of life will evaluate with Nottingham Health Profile, whereas the level of neck disability will evaluate before and after exercise with 'Neck Pain and Disability Score' (NPDS). The obtained results will analyze using appropriate statistical methods.

DETAILED DESCRIPTION:
The treatment program will be applied 3 days a week for 8 weeks.Each 2 groups; will be evaluated twice, at the beginning of the treatment and at the end of the 8th week.

Conventional physiotherapy program consists of neck isometric exercises, neck isotonic exercises, stabilization exercises, stretching exercises and posture exercises and physiotherapy agents.

Neuroscience education; The trainings will be conducted in the form of face-to-face interviews and 45-50 minute one-to-one sessions.

Posters, pictures, graphics and stories, as well as booklets and videos from Explain Pain, Pain in motion and retrainpain websites will be used in appropriate sessions.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-65
* neck pain that persists for 3 months or more

Exclusion Criteria:

* Patients undergoing cervical surgery
* Patients with neck pain secondary to neurological or vascular disease or neoplasia
* Patients with radiculopathy with neurological deficits
* Patients with a history of inflammatory or infective arthritis of the cervical spine
* Patients who received a physical therapy program in the last 6 months
* Patients with pain in the scapula, shoulder, upper extremity or lumbar region that may interfere with neck stabilization exercises

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 8 weeks
  Self reported pain intensity .. Pain intensity was evaluated before and after exercise with 'Visual Analog Scale'. Each item scored is 0-10 (0=no pain 10=pain as bad as can be)
Range Of Motion | 8 weeks
  The CROM (Cervical Range-of-Motion Instrument) combines AMA-required inclinometers and magnets in an easy-to-use instrument. It eliminates positioning, zeroing and tracking errors that are common with stand-alone inclinometers. Standardized protocol minimizes the chance of examination error.
Kinesiofobia | 8 weeks
  Self reported. The Nottingham Health Profile (NHP) was originally created as a standardised tool to survey health problems and measure medical or social interventions. Respondents tick yes or no boxes to answer questions about their health and its effects on their daily life.
Disability | 8 weeks
  Self reported. The level of neck disability was evaluated before and after exercise with 'Neck Pain and Disability Score' . Each question is measured on a scale from 0 (no disability) to 5, and an overall score out of 100 is calculated by adding each item score together.
Quality of life level | 8 weeks
  Self reported. The Nottingham Health Profile (NHP) was originally created as a standardised tool to survey health problems and measure medical or social interventions. Respondents tick yes or no boxes to answer questions about their health and its effects on their daily life.
Pain pressure threshold | 8 weeks
  Algometers are devices that can be used to identify the pressure and/or force eliciting a pressure-pain threshold. It has been noted in pressure-pain threshold studies that the rate at which manual force is applied should be consistent to provide the greatest reliability.
Pain knowledge | 8 weeks
  Self reported. The Neurophysiology of Pain Questionnaire (NPQ) was devised to assess how an individual conceptualizes the biological mechanisms that underpin his or her pain. presents 12 items, and the answer options also consist of "true, false or undecided". Its psychometric properties constitute a one- -dimensional scale with good test-retest reliability. The results are interpreted as follows: each hit corresponds to one point, if the individual makes a mistake or choose the "undecided" alternati- ve, the item is reset to zero; therefore, the score ranges from zero to 12, and the higher the score, the greater the level of unders- tanding of the mechanisms present in pain

CONTACTS AND LOCATIONS:
Locations (1):
- Özden YAŞARER, Istanbul, Turkey (Türkiye)